CLINICAL TRIAL: NCT01048281
Title: Clinical & Pathological Studies of Upper Gastrointestinal Carcinoma
Status: Recruiting | Type: Observational
Sponsor: Stanford University (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Other Study IDs: IRB-13473; 76274 (Other: Stanford University Alternate IRB Approval Number); CA109190 (Other: NIH); SU-11022007-787 (Other: Stanford University)
Record Dates: First submitted 2010-01-11; First posted 2010-01-13 (Estimated); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Stomach Cancer; Gastro-Esophageal(GE) Junction Cancer; Gastric (Stomach) Cancer; Esophageal Cancer; Gastrointestinal Stromal Tumor (GIST)
MeSH Terms: conditions — Stomach Neoplasms; Esophageal Neoplasms; Gastrointestinal Stromal Tumors | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood, tumor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Blood draw
Procedure: Tissue tumor biopsy

SUMMARY:
Our research of the biology of upper gastrointestinal cancers involves the study of tissue samples and cells from biopsies of persons with gastric or esophageal cancer or blood samples from upper gastrointestinal cancer patients and persons at high inherited risk for these cancers. We hope to learn the role genes and proteins play in the development of gastric and esophageal cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Over 18
2. Diagnosed with gastric or esophageal cancer OR at an increased hereditary risk for upper GI cancer

Exclusion Criteria:

1. Under 18
2. No family or personal history of gastric or esophageal cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with gastric or esophageal cancer
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2002-08; Primary Completion 2099-01 (Estimated); Study Completion 2099-01 (Estimated)

PRIMARY OUTCOMES:
p53 activity by routine pathologic analysis | time of collection
NER activity by routine pathologic analysis | time of collection

CONTACTS AND LOCATIONS:
Overall Officials: James M Ford, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States